CLINICAL TRIAL: NCT06737211
Title: Optimizing Postoperative Nutrition in Colorectal Surgery: a Prospective Randomized Clinical Trial.
Brief Title: Optimizing Postoperative Nutrition in Colorectal Surgery
Acronym: OPTI-NUTRICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Maximos Frountzas, Principal Investigator, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPTI-NUTRICS study
Record Dates: First submitted 2024-12-07; First posted 2024-12-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Diseases; Bowel Ischemia; Malnutrition; Parenteral Nutrition
Keywords: peripheral parenteral nutrition; postoperative outcomes; colorectal surgery; colorectal cancer; inflammatory bowel disease; bowel ischemia
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Malnutrition; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 2000 mL of peripheral parenteral nutrition with electrolytes (20 mL 7.45% KCl, 10 mL 20% MgSO4 and 20 mL 8.7% Na3PO4) will be administered via a peripheral venous catheter with a rhythm of 80cc/h from the time they will leave the operation room and will be transferred to the ward or the critical care unit (CCU) until the 5th postoperative day
  Interventions: Dietary Supplement: Peripheral Parenteral Nutrition
- Control (No Intervention): 1000 mL of 10% glucose saline with electrolytes (20 mL 7.45% KCl, 10 mL 20% MgSO4 and 20 mL 8.7% Na3PO4) will be administered via a central or peripheral venous catheter with a rhythm of 80cc/h until the 5th postoperative day

INTERVENTIONS:
Dietary Supplement: Peripheral Parenteral Nutrition — 2000 mL of peripheral parenteral nutrition with electrolytes (20 mL 7.45% KCl, 10 mL 20% MgSO4 and 20 mL 8.7% Na3PO4) will be administered via a peripheral venous catheter with a rhythm of 80cc/h from the time they will leave the operation room and will be transferred to the ward or the critical care unit (CCU) until the 5th postoperative day
  Arms: Intervention

SUMMARY:
Major surgical operations of the gastrointestinal tract, such as colorectal resections due to several diseases, lead to significant burden on the human body, which is expressed during the first postoperative hours with an intense inflammatory reaction and consumption of a large amount of energy, increasing nutritional requirements of the patients. Therefore, specific protocols have been implemented for the early initiation of oral feeding in patients undergoing colorectal resections. However, it is not feasible for every patient to meet them due to several reasons, such as old age and associated pathophysiological changes, use of opioid drugs for the management of postoperative pain, which is associated with postoperative ileus or nausea, as well as open resection which lead to gastrointestinal impairment during the first postoperative days. The energy deficit that occurs during the early postoperative period, which appears to be associated with adverse clinical outcomes, can be counterbalanced by the administration of parenteral nutrition. However, the conventional way of administration through central venous lines is associated with significant complications. For this reason, administration of parenteral nutrition through a peripheral venous catheter could be used alternatively, which avoids morbidity and has been also effective in maintaining the patients' energy balance, even during the first postoperative hours. Therefore, the main purpose of the present study is to investigate the efficacy of the administration of peripheral parenteral nutrition on the postoperative outcomes of patients undergoing colorectal resections. Moreover, the correlation of the administration of peripheral parenteral nutrition with the reaction to post-operative stress and with the nutritional status of the patients post-operatively, which are determining factors for the clinical course of these patients, will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal resection surgery
* Open or laparoscopic procedures
* Anastomosis, end-stoma or defunctioning stoma formation after colorectal resection
* Elective or emergent procedures
* Diagnosis of colorectal cancer, inflammatory bowel disease, diverticular disease and bowel ischemia
* Small bowel resection combined with colorectal resection
* Age > 18 years old
* Informed consent

Exclusion Criteria:

* Small bowel resection without colorectal resection
* End-stoma or defunctioning stoma formation without colorectal resection
* Preoperative parenteral nutrition administration
* Administration of parenteral nutrition after the 4th postoperative day
* Peripheral parenteral nutrition initiation after the 1st postoperative day
* Contraindication for peripheral parenteral nutrition administration
* Age < 18 years old
* No informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Postoperative Surgical Stress and Short-term Nutritional Status | 5 postoperative days
  Serum nutritional markers and acute phase proteins indicating postoperative surgical stress response.

SECONDARY OUTCOMES:
Postoperative Morbidity | 90 postoperative days
  Complications after surgery and their classification according to Calvin-Dindo score.
Nasogastric tube removal | 30 postoperative days
  Postoperative day of nasogastric tube removal
Feeding start | 30 postoperative days
  Postoperative day of feeding start
Early mobilization | 30 postoperative days
  Postoperative day of mobilization
Opioid sparing analgesia | 30 postoperative days
  Utilization of epidural sparing catheter
Peripheral Parenteral Nutrition - associated complications | 30 postoperative days
  Thrombophlebitis, hyperglycemia, re-feeding syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Hippocration General Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Studer P, Raber G, Ott D, Candinas D, Schnuriger B. Risk factors for fatal outcome in surgical patients with postoperative aspiration pneumonia. Int J Surg. 2016 Mar;27:21-25. doi: 10.1016/j.ijsu.2016.01.043. Epub 2016 Jan 20. PMID 26804349
- [Background] Herbert G, Perry R, Andersen HK, Atkinson C, Penfold C, Lewis SJ, Ness AR, Thomas S. Early enteral nutrition within 24 hours of lower gastrointestinal surgery versus later commencement for length of hospital stay and postoperative complications. Cochrane Database Syst Rev. 2019 Jul 22;7(7):CD004080. doi: 10.1002/14651858.CD004080.pub4. PMID 31329285
- [Background] Shin CH, Long DR, McLean D, Grabitz SD, Ladha K, Timm FP, Thevathasan T, Pieretti A, Ferrone C, Hoeft A, Scheeren TWL, Thompson BT, Kurth T, Eikermann M. Effects of Intraoperative Fluid Management on Postoperative Outcomes: A Hospital Registry Study. Ann Surg. 2018 Jun;267(6):1084-1092. doi: 10.1097/SLA.0000000000002220. PMID 28288059
- [Background] Cardinale F, Chinellato I, Caimmi S, Peroni DG, Franceschini F, Miraglia Del Giudice M, Bernardini R. Perioperative period: immunological modifications. Int J Immunopathol Pharmacol. 2011 Jul-Sep;24(3 Suppl):S3-12. doi: 10.1177/03946320110240s302. PMID 22014920
- [Background] Gillis C, Carli F. Promoting Perioperative Metabolic and Nutritional Care. Anesthesiology. 2015 Dec;123(6):1455-72. doi: 10.1097/ALN.0000000000000795. PMID 26248016